CLINICAL TRIAL: NCT05383235
Title: Facial Emotion Recognition in Patients Who Committed Sexual Assault Against Children: an EEG Study
Acronym: EMOREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-A02763-38
Record Dates: First submitted 2022-04-20; First posted 2022-05-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Child Sexual Abuse; Emotion Recognition
Keywords: facial emotion recognition; sexual offenders against children; LPP

STUDY DESIGN:
Intervention Model Description: PATIENTS:
  1. ROUTINE CARE : retrieval of sociodemographic characteristics, medical and psychological assessment, multidisciplinary meeting
  2. RUN-IN PERIOD:
     * Eligibility criteria will be assessed during the multidisciplinary meeting
     * Delivery of the information note
  3. STUDY:
     * Collection of consent form
     * Facial emotion stimuli presentation task with EEG recording and facial emotion recognition task
     * Neuropsychological evaluation
     * Scales + questionnaires
     * Debriefing
  CONTROLS:
  1. RUN-IN PERIOD phone call:
     * Study presentation
     * Retrieval of sociodemographic characteristics including age and educational level for matching with patients
     * Assessment of eligibility criteria
     * Psychiatric assessment with MINI 5.0 evaluation
  2. STUDY:
     * Delivery of the information note
     * Collection of consent form
     * Facial emotion stimuli presentation task with EEG recording and facial emotion recognition task
     * Neuropsychological evaluation
     * Scales + questionnaires
     * Debriefing
Who Masked: Outcomes Assessor
Masking Description: Apart from investigators in charge of inclusions, outcome assessors will not know to which group the subjects belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual offenders against children (Experimental): sexual offenders against children
  Interventions: Other: ROUTINE CARE; Device: Facial emotion stimuli prensentation task with EEG recording and facial emotion recognition task
- Healthy controls (Active Comparator): Healthy controls
  Interventions: Device: Facial emotion stimuli prensentation task with EEG recording and facial emotion recognition task

INTERVENTIONS:
Other: ROUTINE CARE — 1. ROUTINE CARE : retrieval of sociodemographic characteristics, medical and psychological assessment, multidisciplinary meeting about the patient
  Arms: Sexual offenders against children
Device: Facial emotion stimuli prensentation task with EEG recording and facial emotion recognition task — 2. RUN-IN PERIOD :
  * Eligibility criteria will be assessed during the multidisciplinary meeting;
  * Study presentation, delivery of the information note and consent form; 3. STUDY:
  * Collection of consent form;
  * Facial emotion stimuli presentation task with EEG recording and facial emotion recording task;
  * Neuropsychological evaluation (TOM-15);
  * Scales and questionnaires (TAS-20, PCL-R SV, CECAQ, QCAE);
  * Debriefing.
  Other Names: Neuropsychological evaluation

SUMMARY:
This study aims to compare the emotional processing in sexual offenders against children versus healthy volunteers using an objective electrophysiological measurement (EEG) during a facial emotion stimuli presentation task. Secondary goal is to assess emotion recognition performances in this population and evaluate the impact of various factors on these performances (type of emotion, age and sex of person expressing the emotion, neuropsychological and cognitive abilities of the subjects).

DETAILED DESCRIPTION:
Sexual abuse is a major public health issue. Apart from medical care of victims, it appears essential to intervene with sexual offenders for prevention purposes (from primary prevention to avoid a first sexual abuse to secondary and tertiary prevention to avoid recurrence). In order to improve those prevention strategies, further understanding of offenders neuropsychological and cognitive processes is needed.

Facial emotion recognition capacities, that play a major role in social cognition and generation of appropriate social behavior, has been the subject of few studies in sexual offenders. These studies show heterogeneous results and only one of them specifically targets sexual offenders against children. Furthermore, no study has investigated facial emotion recognition in this population with an objective measurement of emotional processing, such as electroencephalographic (EEG) activity. LPP (late positive potential) amplitude, measured in EEG, is a marker of emotional processing and appears to be modified in particular populations (eg. psychopaths) in response to negative visual stimuli compared to positive stimuli.

The investigators aim to determine whether LPP amplitude in response to negative facial expressions is modified in sexual offenders against children compared to healthy volunteers and compared to amplitude in response to positive facial expressions.

Effect of facial emotion characteristics (type of emotion, age and sex of person expressing the emotion) on EEG response will be assessed.

Various neuropsychological and cognitive characteristics (facial emotion recognition, theory of mind, psychopathic traits, childhood trauma, and alexithymia) of patients and controls will also be measured through neuropsychological evaluation and completion of scales and questionnaires, in order to investigate the impact of those factors on facial emotion recognition performances.

ELIGIBILITY:
Inclusion Criteria SUBJECTS - Sexual offenders against children:

* Right-handed ;
* Patient refered to the referral platform for treatment of sexual offenders in Le Vinatier Hospital Center for evaluation of child abuse ;
* Without any Axis 1 disorder ;
* Having given informed consent ;
* Affiliated to French social health care

Exclusion Criteria:

* Intellectual disability (identified during routine care in the referral platform for treatment of sexual offenders);
* Poor understanding of tests and scales instructions ;
* Neurological or neurodevelopmental history resulting in cognitive impairment with loss of autonomy ;
* Gardianship or other tutelage measure

Healthy controls :

Inclusion Criteria:

* Right-handed ;
* Without criminal background ;
* Without any DSM-5 psychiatric disorder (past or present, personal or familial in a first-degree relative) ;
* Non-caregiver employee of Le Vinatier Hospital Center.

Exclusion Criteria:

* Intellectual disability (using fNART if clinical suspicion during run-in period);
* Poor understanding of tests and scales instructions ;
* Neurological or neurodevelopmental history resulting in cognitive impairment with loss of autonomy ;
* Gardianship or other tutelage measure.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Amplitude of LPP during the facial emotion stimuli presentation task | one day
  The facial emotion stimuli presentation task is based on pictures from the Radbout Faces Database (RaFD). It includes pictures of male and female subjects, adults and children expressing positive, neutral or negative emotion.
  During the task, cerebral activity will be recorded by EEG to measure amplitude and latency of the LPP (Late Positive Potential).

SECONDARY OUTCOMES:
Facial emotion recognition abilities | one day
  Subjects and controls will be presented with facial emotion stimuli from the Radbout Faces Database (RaFD). It includes pictures of male and female subjects, adults and children expressing positive, neutral or negative emotion.
  We will measure recognition abilities (% correct response rate, response time, intensity and valence ratings).
TOM-15 (Theory Of Mind 15) | one day
  validated test for assessment of theory of mind
TAS20 (Toronto Alexithymia Scale 20) | one day
  validated scale for assessment of alexithymia Scores vary from 20/100 (low level of alexithymia) to 100/100 (high level of alexithymia)
PCL-R SV (Psychopathy Checklist Revised - Short Version) | one day
  validated checklist for assessment of psychopathy Scores vary from 0/24 (no psychopathic traits) to 24/24 (high level of psychopathic traits)
QCAE (Questionnaire of Cognitive and Affective Empathy) | one day
  validated questionnaire for assessment of cognitive and affective empathy Affective empathy scores vary from 12/48 (low level of affective empathy) to 48/48 (high level of affective empathy).
  Cognitive empathy scores vary from 19/76 (low level of cognitive empathy) to 76/76 (high level of cognitive empathy).
  Total empathy scores vary from 31/124 (low level of empathy) to 124/124 (high level of empathy).
CECA-Q (Childhood Experiences of Care and Abuse - Questionnaire) | one day
  validated questionnaire for assessment of childhood experience of care and abuse Global parental antipathy scores vary from 20/160 (low level of parental antipathy) to 160/160 (high level of parental antipathy).
  Neglect scores vary from 20/160 (low level of neglect) to 160/160 (high level of neglect).
  Physical abuses scores vary from 0/8 (no physical abuses) to 8/8 (high level of physical abuses during childhood) Scores of sexual abuse vary from 0 (no sexual abuse) à 7 (serious sexual abuse) Prevalence of psychological abuse vary from 0/34 (no psychological abuse) to 34/34 (multiple psychological abuses) Frequence of psychological abuse vary from 0/102 ( no psychological abuse) to 102/102 (frequent psychological abuse)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine MOUCHET, PH, Principal Investigator — CH le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No